CLINICAL TRIAL: NCT01848457
Title: Pilot Study to Prevent Nephrotoxicity of High-Dose Methotrexate by Prolonging the Infusion Duration and Prevent Nephrotoxicity and Ototoxicity of Cisplatin With Pantoprazole in Children, Adolescents and Young Adults With Osteosarcoma
Brief Title: Preventing Nephrotoxicity and Ototoxicity From Osteosarcoma Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Gateway for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-009967; CHP12ST051 OS Pilot (Other: The Children's Hospital of Philadelphia)
Record Dates: First submitted 2013-04-29; First posted 2013-05-07 (Estimated); Results first posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Osteosarcoma; Nephrotoxicity; Ototoxicity
Keywords: Osteosarcoma; Cancer; Nephrotoxicity; Ototoxicity; Cisplatin; High-dose methotrexate; Biomarkers; Patient reported outcomes
MeSH Terms: conditions — Osteosarcoma; Ototoxicity; Neoplasms | interventions — Pantoprazole; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cycles 1 & 2: HDMTX 4 h, PTZ+C; Cycles 3 & 4: HDMTX 12 h, C (Experimental): Cycles 1 and 2: HDMTX administered as a 4-hour infusion and pantoprazole is administered with cisplatin Cycles 3 and 4: HDMTX administered as a 12-hour infusion and cisplatin is administered alone
  Interventions: Drug: Pantoprazole; Drug: High-dose methotrexate infusion duration
- Cycles 1 & 2: HDMTX 4 h, C; Cycles 3 & 4: HDMTX 12 h, PTZ + C (Experimental): Cycles 1 and 2: HDMTX administered as a 4-hour infusion and cisplatin is administered alone Cycles 3 and 4: HDMTX administered as a 12-hour infusion and pantoprazole is administered with cisplatin
  Interventions: Drug: Pantoprazole; Drug: High-dose methotrexate infusion duration
- Cycles 1 & 2: HDMTX 12 h, PTZ+C; Cycles 3 & 4: HDMTX 4 h, C (Experimental): Cycles 1 and 2: HDMTX administered as a 12-hour infusion and pantoprazole is administered with cisplatin Cycles 3 and 4: HDMTX administered as a 4-hour infusion and cisplatin is administered alone
  Interventions: Drug: Pantoprazole; Drug: High-dose methotrexate infusion duration
- Cycles 1 & 2: HDMTX 12 h, C; Cycles 3 & 4: HDMTX 4 h, C + PTZ (Experimental): Cycles 1 and 2: HDMTX administered as a 12-hour infusion and cisplatin is administered alone Cycles 3 and 4: HDMTX administered as a 4-hour infusion and pantoprazole is administered with cisplatin
  Interventions: Drug: Pantoprazole; Drug: High-dose methotrexate infusion duration

INTERVENTIONS:
Drug: Pantoprazole — 0.3 mg/kg IV over 15 min immediately prior to cisplatin as a loading dose on days 1 & 2 followed by 1.3 mg/kg IV infused over 4 h concurrent with the 4 h cisplatin infusion on days 1 & 2 of treatment Cycles 1 & 2 (Treatment Arms 1, 3) OR Cycles 3 & 4 (Treatment Arms 2, 4)
  Other Names: Protonix IV
Drug: High-dose methotrexate infusion duration — High-dose methotrexate (12 g/sq m, maximum dose 20 g) will be infused over 4 hours or 12 hours
  Other Names: Otrexup (PF), Xatmep, Trexall

SUMMARY:
Osteosarcoma is the most common type of bone cancer in children, adolescents and young adults. Treatment with surgery and a combination of three conventional chemotherapy drugs can cure nearly two-thirds patients with osteosarcoma, but the treatment can also cause irreversible damage to the kidneys and cause permanent hearing loss. The purpose of this study is to evaluate new approaches to prevent these side effects without interfering with the beneficial effects of the chemotherapy drugs on the cancer by using our knowledge of how the drugs damage the kidney and cochlear hair cells in the ear to selectively block these side effects. Preventing these side effects without interfering with the anti-cancer effect of the drugs will improve the outcome in survivors and may also improve the effectiveness of the chemotherapy regimen by preventing treatment delays and dose reductions that are often caused by the side effects. Patients will be carefully monitored to ensure that the new interventions do not adversely affect response to the treatment and do not increase the other side effects of the chemotherapy. Specifically, we will monitor the nutritional status of the patients closely and ask patients to complete a survey describing the side effects after each treatment cycle. We will also collect a small sample of cancer tissue at the time of biopsy and surgery from each patient on this study for testing to determine new classes of anti-cancer drugs currently under development may have a role in treating osteosarcoma. If effective, these new approaches to prevent kidney damage and hearing loss will be applicable in other types of cancers treated with the same chemotherapy drugs.

DETAILED DESCRIPTION:
Current osteosarcoma treatment regimens include cisplatin and high-dose methotrexate (HDMTX), which are nephrotoxic and ototoxic, and the damage to kidneys and cochlear hair cells may be irreversible. Preventing these toxicities will improve the outcome in long-term survivors and may also prevent short-term treatment delays and dose reductions that can compromise the efficacy of the treatment regimen and allow for administration of higher cumulative doses of cisplatin. This pilot study evaluates pharmacologically-based approaches to prevent the nephrotoxic effect of HDMTX by prolonging the infusion duration and thereby lowering the risk of drug precipitation in renal tubules; and to selectively block the uptake of cisplatin into renal tubular cells and cochlear hair cells by inhibiting the organic cation transporter 2 (OCT2) with the proton pump inhibitor (PPI), pantoprazole. Participants with previously untreated biopsy-proven, localized or metastatic osteosarcoma will receive six cycles of the standard Methotrexate, Adriamycin (doxorubicin),cisplatin (MAP) chemotherapy regimen, which includes high-dose methotrexate, doxorubicin and cisplatin. The first 2 cycles are administered neoadjuvantly followed by surgery to remove the primary tumor, when feasible.

A novel randomized, crossover, 2 x 2 factorial clinical trial design allows all patients to receive the new interventions to prevent toxicity and to serve as their own controls. New, sensitive urinary biomarkers of acute kidney injury serve as primary endpoints for evaluating treatment-related renal damage. Ototoxicity will be monitored using audiograms. The effect of these interventions on tumor response (radiographic and histologic) and toxicity (including a patient reported outcome survey and nutritional status) will be closely monitored. Other secondary objectives include evaluating bone-specific alkaline phosphatase as a biomarker of tumor burden and constructing a tissue microarray to evaluate expression of proteins that are responsible for resistance to the current drugs used to treat osteosarcoma and assess expression of proteins that are targeted by new anticancer drugs under development for childhood cancers.

ELIGIBILITY:
Inclusion Criteria:

* <30 years of age
* histological diagnosis of high-grade osteosarcoma
* Extremity or central axis (including craniofacial) primary tumor; localized or metastatic
* No prior chemotherapy or radiation therapy for osteosarcoma. Subjects who develop osteosarcoma as a second cancer are eligible if they have not previously received cisplatin, doxorubicin or other anthracyclines, or MTX
* Serum creatinine at or below the upper limit of normal (ULN) for age and gender
* Shortening fraction on echocardiogram >28%
* Hearing level threshold ≤25 dB at all frequencies in both ears to be evaluable for evaluation of pantoprazole's effect on cisplatin ototoxicity. Patients with hearing loss can be enrolled but will not be evaluable for ototoxicity objective.
* Absolute neutrophil count >1,000/microliter(mcL) and platelet count >100,000/mcL

Exclusion Criteria:

* Receiving H2 antagonists (cimetidine, ranitidine, famotidine, nizatidine) or proton pump inhibitors (lansoprazole, omeprazole, pantoprazole, esomeprazole, rabeprazole, dexlansoprazole) AND unable to hold the drug for 24 h prior to and 24 h after each cisplatin course on cycles 1-4.
* Pregnant or breastfeeding
* Unable to cooperate with research procedures

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2016-01-04 (Actual); Study Completion 2016-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank M Balis, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Fox E, Busch C, DeBernardo A, Segers B, Gottschalk J, Womer R, Balamuth N, Bagatell R, Balis F. A pharmacologically-based approach to high dose methotrexate administration to investigate nephrotoxicity and acute kidney injury biomarkers in children and adolescents with newly diagnosed osteosarcoma. Cancer Chemother Pharmacol. 2021 Jun;87(6):807-815. doi: 10.1007/s00280-021-04248-8. Epub 2021 Mar 7. PMID 33677616
- [Derived] Fox E, Levin K, Zhu Y, Segers B, Balamuth N, Womer R, Bagatell R, Balis F. Pantoprazole, an Inhibitor of the Organic Cation Transporter 2, Does Not Ameliorate Cisplatin-Related Ototoxicity or Nephrotoxicity in Children and Adolescents with Newly Diagnosed Osteosarcoma Treated with Methotrexate, Doxorubicin, and Cisplatin. Oncologist. 2018 Jul;23(7):762-e79. doi: 10.1634/theoncologist.2018-0037. Epub 2018 Feb 14. PMID 29445029

RESULTS

PARTICIPANT FLOW:
Groups:
- Cycles 1 & 2: HDMTX 4h, PTZ+C; Then Cycles 3 & 4: HDTMX 12h, C: Cycles 1 and 2: HDMTX administered as a 4-hour infusion and pantoprazole is administered with cisplatin Cycles 3 and 4: HDMTX administered as a 12-hour infusion and cisplatin is administered alone
  Pantoprazole: 0.3 mg/kg IV over 15 min immediately prior to cisplatin as a loading dose on days 1 & 2 followed by 1.3 mg/kg IV infused over 4 h concurrent with the 4 h cisplatin infusion on days 1 & 2 of treatment Cycles 1 & 2 (Treatment Arms 1, 3) OR Cycles 3 & 4 (Treatment Arms 2, 4)
  High-dose methotrexate infusion duration: High-dose methotrexate (12 g/sq m, maximum dose 20 g) will be infused over 4 hours or 12 hours
- Cycles 1 & 2: HDMTX 4h, C; Then Cycles 3 & 4: HDTMX 12h, C+PTZ: Cycles 1 and 2: HDMTX administered as a 4-hour infusion and cisplatin is administered alone Cycles 3 and 4: HDMTX administered as a 12-hour infusion and pantoprazole is administered with cisplatin
  Pantoprazole: 0.3 mg/kg IV over 15 min immediately prior to cisplatin as a loading dose on days 1 & 2 followed by 1.3 mg/kg IV infused over 4 h concurrent with the 4 h cisplatin infusion on days 1 & 2 of treatment Cycles 1 & 2 (Treatment Arms 1, 3) OR Cycles 3 & 4 (Treatment Arms 2, 4)
  High-dose methotrexate infusion duration: High-dose methotrexate (12 g/sq m, maximum dose 20 g) will be infused over 4 hours or 12 hours
- Cycles 1 & 2: HDMTX 12h, PTZ+C; Then Cycles 3 & 4: HDTMX 4h, C: Cycles 1 and 2: HDMTX administered as a 12-hour infusion and pantoprazole is administered with cisplatin Cycles 3 and 4: HDMTX administered as a 4-hour infusion and cisplatin is administered alone
  Pantoprazole: 0.3 mg/kg IV over 15 min immediately prior to cisplatin as a loading dose on days 1 & 2 followed by 1.3 mg/kg IV infused over 4 h concurrent with the 4 h cisplatin infusion on days 1 & 2 of treatment Cycles 1 & 2 (Treatment Arms 1, 3) OR Cycles 3 & 4 (Treatment Arms 2, 4)
  High-dose methotrexate infusion duration: High-dose methotrexate (12 g/sq m, maximum dose 20 g) will be infused over 4 hours or 12 hours
- Cycles 1 & 2: HDMTX 12h, C; Then Cycles 3 & 4: HDTMX 4h, C+PTZ: Cycles 1 and 2: HDMTX administered as a 12-hour infusion and cisplatin is administered alone Cycles 3 and 4: HDMTX administered as a 4-hour infusion and pantoprazole is administered with cisplatin
  Pantoprazole: 0.3 mg/kg IV over 15 min immediately prior to cisplatin as a loading dose on days 1 & 2 followed by 1.3 mg/kg IV infused over 4 h concurrent with the 4 h cisplatin infusion on days 1 & 2 of treatment Cycles 1 & 2 (Treatment Arms 1, 3) OR Cycles 3 & 4 (Treatment Arms 2, 4)
  High-dose methotrexate infusion duration: High-dose methotrexate (12 g/sq m, maximum dose 20 g) will be infused over 4 hours or 12 hours
Period: Overall Study
Arm/Group | Cycles 1 & 2: HDMTX 4h, PTZ+C; Then Cycles 3 & 4: HDTMX 12h, C | Cycles 1 & 2: HDMTX 4h, C; Then Cycles 3 & 4: HDTMX 12h, C+PTZ | Cycles 1 & 2: HDMTX 12h, PTZ+C; Then Cycles 3 & 4: HDTMX 4h, C | Cycles 1 & 2: HDMTX 12h, C; Then Cycles 3 & 4: HDTMX 4h, C+PTZ
Started | 4 | 3 | 3 | 3
Baseline | 4 | 3 | 3 | 3
Cycle 1 | 4 | 3 | 3 | 3
Cycle 2 | 3 | 3 | 3 | 3
Cycle 3 | 3 | 3 | 3 | 3
Cycle 4 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 1 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Cycles 1 and 2: HDMTX administered as a 4-hour infusion and pantoprazole is administered with cisplatin Cycles 3 and 4: HDMTX administered as a 12-hour infusion and cisplatin is administered alone
  Pantoprazole: 0.3 mg/kg IV over 15 min immediately prior to cisplatin as a loading dose on days 1 & 2 followed by 1.3 mg/kg IV infused over 4 h concurrent with the 4 h cisplatin infusion on days 1 & 2 of treatment Cycles 1 & 2 (Treatment Arms 1, 3) OR Cycles 3 & 4 (Treatment Arms 2, 4)
  High-dose methotrexate infusion duration: High-dose methotrexate (12 g/sq m, maximum dose 20 g) will be infused over 4 hours or 12 hours
- Arm 2: Cycles 1 and 2: HDMTX administered as a 4-hour infusion and cisplatin is administered alone Cycles 3 and 4: HDMTX administered as a 12-hour infusion and pantoprazole is administered with cisplatin
  Pantoprazole: 0.3 mg/kg IV over 15 min immediately prior to cisplatin as a loading dose on days 1 & 2 followed by 1.3 mg/kg IV infused over 4 h concurrent with the 4 h cisplatin infusion on days 1 & 2 of treatment Cycles 1 & 2 (Treatment Arms 1, 3) OR Cycles 3 & 4 (Treatment Arms 2, 4)
  High-dose methotrexate infusion duration: High-dose methotrexate (12 g/sq m, maximum dose 20 g) will be infused over 4 hours or 12 hours
- Arm 3: Cycles 1 and 2: HDMTX administered as a 12-hour infusion and pantoprazole is administered with cisplatin Cycles 3 and 4: HDMTX administered as a 4-hour infusion and cisplatin is administered alone
  Pantoprazole: 0.3 mg/kg IV over 15 min immediately prior to cisplatin as a loading dose on days 1 & 2 followed by 1.3 mg/kg IV infused over 4 h concurrent with the 4 h cisplatin infusion on days 1 & 2 of treatment Cycles 1 & 2 (Treatment Arms 1, 3) OR Cycles 3 & 4 (Treatment Arms 2, 4)
  High-dose methotrexate infusion duration: High-dose methotrexate (12 g/sq m, maximum dose 20 g) will be infused over 4 hours or 12 hours
- Arm 4: Cycles 1 and 2: HDMTX administered as a 12-hour infusion and cisplatin is administered alone Cycles 3 and 4: HDMTX administered as a 4-hour infusion and pantoprazole is administered with cisplatin
  Pantoprazole: 0.3 mg/kg IV over 15 min immediately prior to cisplatin as a loading dose on days 1 & 2 followed by 1.3 mg/kg IV infused over 4 h concurrent with the 4 h cisplatin infusion on days 1 & 2 of treatment Cycles 1 & 2 (Treatment Arms 1, 3) OR Cycles 3 & 4 (Treatment Arms 2, 4)
  High-dose methotrexate infusion duration: High-dose methotrexate (12 g/sq m, maximum dose 20 g) will be infused over 4 hours or 12 hours
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Total
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 3 | 2 | 3 | 12
  Between 18 and 65 years | 0 | 0 | 1 | 0 | 1
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 14.3 [9 to 17] | 10.3 [5 to 17] | 8.3 [6 to 19] | 10.7 [7 to 14] | 11.4 [5 to 19]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 1 | 8
  Male | 2 | 0 | 1 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 3 | 3 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 3 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in Urinary Biomarkers of Acute Kidney Injury (AKI) Between Pre-Treatment (Baseline), After CISplatin (C) Treatments, and After HDTMX Treatments
Description: This measure describes the urinary biomarkers of AKI after each course of C throughout Cycles 1-2, compared to baseline (pre-infusion) values.
  Biomarkers of AKI, include: Kidney Injury Molecule-1 (KIM-1), and Neutrophil Gelatinase-Associated Lipocalin (NGAL).
Time Frame: Pretreatment/Baseline, Day 2 of Cycles 1 & 2, Day 8 of Cycles 1 & 2
Population: The original treatment arms/groups are paired down by the arms that include PTZ in the CISplatin infusions, and the arms that do not include PTZ in the CISplatin infusions. This is a general comparison of the changes in AKI measurements when using the PTZ inhibitor, whether HDTMX is infused for 4 or 12 hours.
Measure: Median (Full Range); unit: μg/g
Groups:
- Treatments Arms 1 & 3 (Groups With PTZ in Cycles 1 & 2): Arm 1 receives a 4-hour infusion of HDTX, and Arm 3 receives a 12-hour infusion of HDTMX, during Cycles 1 & 2. Both arms also receive C and PTZ during Cycles 1 & 2.
- Treatments Arms 2 & 4 (Groups Without PTZ in Cycles 1 & 2): Am 2 receives a 4-hour infusion of HDTMX, and Arm 4 receives a 12-hour infusion of HDTMX during Cycles 1 & 2. Both arms also receive the C doses, but without PTZ.
Arm/Group | Treatments Arms 1 & 3 (Groups With PTZ in Cycles 1 & 2) | Treatments Arms 2 & 4 (Groups Without PTZ in Cycles 1 & 2)
Number analyzed (Participants) | 6 | 6
μg/g
  Day 1 Kim-1 (Pretreatment) | 1.7 [0.5 to 5.9] | 1.7 [0.3 to 15]
  Day 2 Kim-1 (post 2 doses Cisplatin) | 2.1 [0.2 to 182] | 3.3 [0.2 to 8.1]
  Day 8 Kim-1 (post HDTMX infusion) | 4.1 [0.5 to 11] | 4.6 [0.4 to 11]
  Day 1 NGAL (Pretreatment) | 18 [2 to 900] | 10 [2.9 to 165]
  Day 2 NGAL (post 2 doses Cisplatin) | 27 [2.6 to 542] | 18 [1.1 to 209]
  Day 8 NGAL (post HDTMX infusion) | 12 [2.2 to 1193] | 12 [1.6 to 841]

2. Secondary Outcome: Change in Tumor Volume
Description: Response of the primary tumor to the first two treatment cycles (Cycles 1 and 2) will be assessed by quantifying the change in tumor volume on MRI, after treatment (pre-operative) relative to the pre-treatment tumor volume. By using the log ratio of the tumor volume post-treatment, to the tumor volume pre-treatment. The larger the change, the more effective the treatment.
Time Frame: Baseline (Week 1), Pre-operative (Month 2)
Measure: Count of Participants; unit: Participants
Groups:
- Localized Disease at Baseline: Cycles 1 and 2: HDMTX administered as a 4-hour infusion and pantoprazole is administered with cisplatin Cycles 3 and 4: HDMTX administered as a 12-hour infusion and cisplatin is administered alone
  Pantoprazole: 0.3 mg/kg IV over 15 min immediately prior to cisplatin as a loading dose on days 1 & 2 followed by 1.3 mg/kg IV infused over 4 h concurrent with the 4 h cisplatin infusion on days 1 & 2 of treatment Cycles 1 & 2 (Treatment Arms 1, 3) OR Cycles 3 & 4 (Treatment Arms 2, 4)
  High-dose methotrexate infusion duration: High-dose methotrexate (12 g/sq m, maximum dose 20 g) will be infused over 4 hours or 12 hours
- Metastatic Disease at Baseline: Cycles 1 and 2: HDMTX administered as a 12-hour infusion and pantoprazole is administered with cisplatin Cycles 3 and 4: HDMTX administered as a 4-hour infusion and cisplatin is administered alone
  Pantoprazole: 0.3 mg/kg IV over 15 min immediately prior to cisplatin as a loading dose on days 1 & 2 followed by 1.3 mg/kg IV infused over 4 h concurrent with the 4 h cisplatin infusion on days 1 & 2 of treatment Cycles 1 & 2 (Treatment Arms 1, 3) OR Cycles 3 & 4 (Treatment Arms 2, 4)
  High-dose methotrexate infusion duration: High-dose methotrexate (12 g/sq m, maximum dose 20 g) will be infused over 4 hours or 12 hours
Arm/Group | Localized Disease at Baseline | Metastatic Disease at Baseline
Number analyzed (Participants) | 9 | 4
Participants
  Complete Response to Chemotherapy | 9 | 0
  Progressive Disease after Chemotherapy | 0 | 4

3. Secondary Outcome: Validating Urinary Biomarkers
Description: Urinary biomarkers of acute kidney injury (AKI) and glomerular filtration rate (GFR) estimated from serum cystatin C will be compared to standard measures of renal function (serum creatinine, urinalysis, estimated creatinine clearance, fractional excretion of Mg). Single reported values are averaged and reported with full ranges.
Time Frame: Day 1 (Pretreatment/Baseline), Day 8, and Day 22 of Cycles 1 & 2
Measure: Median (Full Range); unit: mL/min per 1.73m2
Groups:
- Treatment Arms 1, 3 (w/ Pantoprazole); Treatment Arms 2, 4 (w/o Pantoprazole): Cycles 1 and 2: HDMTX administered as a 12-hour infusion and cisplatin is administered alone Cycles 3 and 4: HDMTX administered as a 4-hour infusion and pantoprazole is administered with cisplatin
  Pantoprazole: 0.3 mg/kg IV over 15 min immediately prior to cisplatin as a loading dose on days 1 & 2 followed by 1.3 mg/kg IV infused over 4 h concurrent with the 4 h cisplatin infusion on days 1 & 2 of treatment Cycles 1 & 2 (Treatment Arms 1, 3) OR Cycles 3 & 4 (Treatment Arms 2, 4)
  High-dose methotrexate infusion duration: High-dose methotrexate (12 g/sq m, maximum dose 20 g) will be infused over 4 hours or 12 hours
Arm/Group | Treatment Arms 1, 3 (w/ Pantoprazole) | Treatment Arms 2, 4 (w/o Pantoprazole)
Number analyzed (Participants) | 6 | 6
mL/min per 1.73m2
  Day 1 GFRcr (pretreatment) | 131 [96 to 252] | 132 [95 to 252]
  Day 8 GFRcr | 120 [81 to 252] | 124 [81 to 252]
  Day 22 GFRcr | 134 [96 to 252] | 141 [64 to 252]
  Day 1 GFRcysC (pretreatment) | 126 [89 to 169] | 120 [87 to 180]
  Day 8 GFRcysC | 105 [78 to 193] | 109 [72 to 186]
  Day 22 GFRcysC | 122 [94 to 160] | 125 [77 to 176]

4. Secondary Outcome: Tissue Microarray
Description: Tissue microarray will be constructed from biopsy specimens, primary resection and resected metastatic tumors to evaluate the expression of proteins that are responsible for resistance to the drugs in the MAP regimen and to assess expression of proteins that are targeted by new anticancer drugs under development for childhood cancers.
Time Frame: Pretreatment (biopsy) at baseline and postoperative (in between cycle 2 and cycle 3)
Population: The study was completed early and biopsy specimens were not submitted for tissue microarray analysis for any patients.
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Bone Specific Alkaline Phosphatase (BSAP)
Description: Serum BSAP will be longitudinally evaluated as a potential biomarker for osteosarcoma
Time Frame: Pretreatment/Baseline, Cycle 3
Measure: Mean (Full Range); unit: U/L
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 2 | 3 | 3 | 3
U/L
  Pretreatment (baseline) | 197.1 [40.2 to 354] | 265 [106 to 557] | 169.67 [111 to 265] | 179.63 [66.7 to 398]
  Cycle 3 | 73.05 [46.1 to 100] | 106.87 [18.6 to 193] | 71.2 [26.1 to 137] | 76.1 [44.6 to 125]

6. Secondary Outcome: Nutritional Status
Description: Nutritional status (weight, arm circumference, skin fold thickness, pre-albumin) will be throughout the course of treatment
Time Frame: Prior to each cycle (Day 1 of cycles 1-6) and end of therapy (at the end of cycle 6)
Population: The nutritional information collected was not able to be reported, due to the metabolized nature of the data. The data points were not able to be included, because they were not able to be read.
Arm/Group | Individual Subjects
Number analyzed (Participants) | 0

7. Secondary Outcome: Patient Reported Outcome Survey (PROS)
Description: PROS survey measures quality of life for pediatric oncology patients, in 17 scaled questions. Each question scaled 0-4 (0 = Never, 1 = Rarely, 2 = Sometimes, 3 = Often, 4 = Almost Always). The higher the final sum of the questions, the lower the quality of life/more severe the side effects of oncology treatment. Total scores can range between 0 = highest quality of life, and 100 = experiencing most severe side effects of oncology treatment/worst quality of life experience.
Time Frame: Baseline, Cycle 2, Surgery, Cycle 3, Cycle 4, Cycle 5, Cycle 6, and End of Therapy
Population: The number analyzed differed between rows and from the overall number of analyzed subjects, because not all subjects completed PROS questionnaires during study visits due to time limitations, and/or activities of the study procedures.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- All Study Participants (Arms 1-4): All participants in the study, regardless of which arm or order they were randomized to receive the study treatment.
Arm/Group | All Study Participants (Arms 1-4)
Number analyzed (Participants) | 8
score on a scale
  Baseline | 23 [16 to 43]
  Cycle 2 | 30 [17 to 46]
  Surgery: number analyzed (Participants) | 5
  Surgery | 22 [10 to 30]
  Cycle 3: number analyzed (Participants) | 4
  Cycle 3 | 24 [4 to 34]
  Cycle 4: number analyzed (Participants) | 6
  Cycle 4 | 24 [7 to 42]
  Cycle 5: number analyzed (Participants) | 5
  Cycle 5 | 19 [9 to 32]
  Cycle 6: number analyzed (Participants) | 4
  Cycle 6 | 20 [5 to 32]
  End of Therapy: number analyzed (Participants) | 4
  End of Therapy | 17 [12 to 23]

8. Secondary Outcome: Ototoxicity
Description: Average hearing level (HL) threshold in decibels (dB) over the frequency range of 4,000-8,000 hertz (Hz) will be derived separately for each ear from audiograms performed before each dose of cisplatin.
Time Frame: Baseline (Week 1), Day 1 of Cycle 1 (Week 1), Day 1 of Cycle 2(Week 6), Day 1 of Cycle 3(Week 11), Day 1 of Cycle 4 (Week 16), and end of therapy/after the end of cycle 6 (Day 28 of cycle 6, Week 28)
Measure: Mean (Full Range); unit: decibels
Arm/Group | Treatment Arms 1, 3 (w/ Pantoprazole) | Treatment Arms 2, 4 (w/o Pantoprazole)
Number analyzed (Participants) | 7 | 5
decibels
  Baseline Right Ear | 3.6 [0.0 to 8.3] | 3.8 [1.7 to 6.7]
  Baseline Left Ear | 3.3 [0.0 to 5.0] | 5.4 [1.7 to 10]
  End of Therapy Right Ear | 34.6 [11.7 to 58.3] | 26.7 [10 to 41.7]
  End of Therapy Left Ear | 35.0 [23.3 to 58.3] | 26.7 [10 to 41.7]

ADVERSE EVENTS:
Time Frame: Adverse events are tracked from the time of the first subject's enrollment, until completion of study therapy of the last enrolled subject, spanning 3.5 years. Each treatment cycle is 4-5 weeks, and there are 6 treatment cycles per subject (24-30 weeks of treatment cycles). In addition, surgery recovery after Cycle 2 is 1-2 weeks. Each fully evaluable subject participated in the study 25-32 weeks (6-8 months).
Description: Adverse events were tracked according to arms/groups of studies, and the cycles at which they occured for each arm/group. Given the nature of how the interventions were implemented, separating each treatment or intervention would not account for the cause of the adverse event, nor identify the time at which the adverse event occured. In order to be consistent, adverse events are reported according to the arm in which they occured.
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
All-Cause Mortality (participants affected / at risk) | 1/4 | 1/3 | 1/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-04-02): https://cdn.clinicaltrials.gov/large-docs/57/NCT01848457/Prot_SAP_000.pdf